CLINICAL TRIAL: NCT06629584
Title: Phase II Study of Asciminib for Second-line Treatment of Chronic Phase Chronic Myeloid Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0396; NCI-2024-07923 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-09-25; First posted 2024-10-08 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-08

CONDITIONS: Malignant Solid Tumors
MeSH Terms: interventions — asciminib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Asciminib (Experimental): Patients will receive asciminib 80 mg once daily continuously for 28-day cycles for 2 years.
  Interventions: Drug: Asciminib

INTERVENTIONS:
Drug: Asciminib — Patients will receive asciminib 80 mg PO once daily continuously for 28-day cycles for 2 years.

SUMMARY:
This is an open label, phase 2 study investigating asciminib in patients previously treated with one line of TKI therapy.

DETAILED DESCRIPTION:
Primary Objectives:

1. To determine the rate of major molecular response (MMR) at 12 months.

Secondary Objectives:

1. To estimate the proportion of patients achieving a complete cytogenetic response (CCyR), major molecular response (MMR) and molecular response 4 and MR4.5 (MR4.5) by 3, 6, 12 (except for MMR as primary endpoint), 18 and 24 months.
2. To estimate the time to CCyR, MMR, MR4.0 and MR4.5.
3. To determine the safety and tolerability profile of asciminib in the second line setting.
4. To determine the event-free survival (EFS), survival free from transformation to accelerated and blast phase (TFS), and overall survival (OS).
5. To evaluate the rate of adverse events (AEs)

Exploratory Objectives:

1. To describe patient reported outcomes using the MDASI-CML instrument
2. To evaluate development of resistance mutations and their impact on outcomes

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Diagnosis of Ph-positive (by cytogenetics or FISH) or BCR-ABL-positive (by PCR) CML in chronic phase and have received one prior line of therapy with a TKI.
3. History of treatment failure defined as either:

   * BCR::ABL1 >0.1% for patients with intolerance to first-line TKI
   * Less than complete hematologic response (CHR) at ≥3 months
   * No partial cytogenetic response at ≥3 months
   * BCR::ABL1 ≥ 10% at if 3-6 months
   * BCR::ABL1 ≥ 1% at ≥6 months
   * Loss of CCyR or development of mutations or other clonal chromosomal abnormalities at any time during TKI treatment
4. ECOG performance status ≤ 2.
5. Adequate end organ function within 12 days before the first dose of asciminib treatment. Patients with mild to moderate renal and hepatic impairment are eligible if:

   * Total bilirubin ≤ 3.0 x ULN without AST/ALT increase
   * Aspartate transaminase (AST) ≤ 5.0 x ULN
   * Alanine transaminase (ALT) ≤ 5.0 x ULN
   * Serum lipase ≤ 1.5 x ULN. For serum lipase > ULN and ≤ 1.5 x ULN, value should be considered not clinically significant and not associated with risk factors for acute pancreatitis
   * Alkaline phosphatase ≤ 2.5 x ULN
   * Creatinine clearance ≥ 30 mL/min as calculated using Cockcroft-Gault formula
6. The effects of Asciminib on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Women of child-bearing potential must agree to use highly effective methods of contraception during dosing and for 30 days after study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Allowable methods of birth control:

   * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
   * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before the start of study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
   * Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that subject.
   * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
   * Sexually active males must use a condom during intercourse while taking the drug and for 30 days after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

Exclusion Criteria:

1. Patients with a history of T315I mutation.
2. Patients with New York Heart Association (NYHA) Class III or IV congestive heart failure or LVEF < 40% by echocardiogram or multi-gated acquisition (MUGA) scan.
3. Patients with a history of myocardial infarction within the last 6 months or unstable/uncontrolled angina pectoris or history of severe and/or uncontrolled ventricular arrhythmias. Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g., bifascicular block, Mobitz type II and third-degree AV block).
4. Corrected QT interval (QTc) of > 450 milliseconds (ms) on baseline electrocardiogram (ECG or EKG) (using the Fridericia Formula)
5. Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:

   * Risk factors for Torsades de Pointes (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia.
   * Concomitant medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointes that cannot be discontinued or replaced 7 days prior to starting study drug by safe alternative medication.
6. Patients with known active infection with human immunodeficiency virus (HIV) or Hepatitis B or C.
7. Patients with known conditions that would significantly affect the ingestion or gastrointestinal absorption of drugs administered orally.
8. Nursing women, women of childbearing potential (WOCBP) with positive blood or urine pregnancy test, or women of childbearing potential who are not willing to maintain adequate contraception (see inclusion criteria 8)
9. History of acute pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis.
10. ANC < 500/mm3, platelet count < 50,000 mm3.
11. History of other active malignancy within 2 years prior to study entry except for previous or concomitant basal cell skin cancer and previous carcinoma in situ treated curatively.
12. Subject has any other significant medical or psychiatric history that in the opinion of the investigator would adversely affect participation in this study.

Patients should have discontinued therapy with imatinib, bosutinib, dasatinib or nilotinib or other anti-leukemia therapy (except hydroxyurea), at least 48 hours prior to start of study therapy and recovered from any toxicity due to these therapies to at least grade 1. The use of hydroxyurea is allowed immediately prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Major molecular response (MMR) rate by 12 months | at 12 months of therapy
  MMR rate at 12 months with the 95% confidence interval will also be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Ghayas Issa, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org